CLINICAL TRIAL: NCT03141424
Title: Periostin-guided Withdrawal of Inhaled Corticosteroids in Patients With Non-eosinophilic Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Christiane Mosbech, MD, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Asthmaperiostin
Record Dates: First submitted 2017-05-03; First posted 2017-05-05 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Therapeutics; Budesonide; Mometasone Furoate; Beclomethasone; ciclesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (No Intervention): Usual care. Unchanged asthma medication during the entire study period.
- Group B (Experimental): Tapering of ICS over 8 weeks. Dosis reduction of 50% in ICS treatment for 8 weeks, followed by total ICS removal. Other inhaled asthma medication remains unchanged during the entire study period.
  Interventions: Drug: Tapering of inhaled corticosteroid (ICS) treatment

INTERVENTIONS:
Drug: Tapering of inhaled corticosteroid (ICS) treatment — Tapering of ICS treatment over 8 weeks. Follow-up over 52 weeks in total. Dosis reduction of 50% in ICS treatment for 8 weeks, followed by total ICS removal. Other inhaled asthma medication remains unchanged during the entire study period.
  Other Names: budesonide; fluticasone proprionate; mometasone furoate; beclometasone dipropionate; ciclesonide
  Arms: Group B

SUMMARY:
Background: Asthma is a common chronic condition characterized by respiratory symptoms and hyperresponsive airways. According to treatment guidelines, patients with persistent asthma require daily treatment with inhaled corticosteroids (ICS). However, certain subgroups of asthma patients such as non-eosinophilic asthma patients do not respond well to the ICS treatment. In the present study, asthma patients treated with ICS and exhibiting low levels of eosinophilic biomarkers such as S-periostin, FeNO and blood eosinophils, are randomized 1:1 to either 1) tapering of ICS or 2) usual care. Thus, the aim of the present study is to investigate whether patients with non-eosinophilic asthma can sustain their level of disease control during ICS tapering.

Design: This is a randomized, controlled, one-center, non-inferiority study of ICS tapering in patients with non-eosinophilic asthma.

Inclusion and exclusion criteria: 1) Objectively secured asthma diagnosis, 2) Age 18-65 years, 3) ICS treatment equivalent to Budesonide 800 microg daily or more with at least 80% adherence, 4) Serum-periostin < 50 ng/ml, 5) FeNO<25 ppb at all prior visits, 6) Blood-eosinophils<0.15 at screening, 7) no allergic asthma history, 8) no daily smoking within 6 months, 9) no other respiratory disease, 10) no daily treatment with immunosuppressives, 11) no pregnancy, and 12) no history of drug or alcohol abuse.

Endpoints: Primary: Change in Control Questionnaire (ACQ) from baseline to post-tapered ICS and time from baseline to drop-out. Secondary: Change in FeNO, change in Serum-Periostin, change in FEV1, change in blood-eosinophils.

Methods: Relevant patients will be recruited from Respiratory Outpatient Wards. In total, 110 patients will be required. Visits will be performed at screening, at week 0, 4, 8, 12, 16, 26, 52. In the active arm, ICS dosage will be reduced to 50% at week 0 and removed at week 8. All visits include ACQ, FeNO, spirometry, blood eosinophils. S-periostin will be measured at screening and at week 8 and 16.

ELIGIBILITY:
Inclusion Criteria:

* Astma patients followed in the Respiratory Outpatient Ward, Hvidovre Hospital, Amager Hospital or Glostrup Hospital.
* At least one of the following test suggestive for asthma, performed at any time during the outpatient course: 1) FEV1-reversibility on at least 12% and 200 ml after administration of bronchodilator or Prednisolon course, 2) positive bronchial provocation test, such as mannitol, 3) peakflow (PF)-variation of at least 20% assessed during a 14-day period, measured twice daily and at asthmatic symptoms, or 4) Variability in FEV1 on at least 12% and 200 ml
* Age 18-65 years
* Treated with ICS daily in doses equivalent to Budesonide 800 microg daily or more
* ICS adherence of at least 80% during the last year, assessed from used prescriptions
* Serum-periostin < 50 ng/ml at screening (8)
* FeNO < 25 ppb at all prior visits
* Blood-eosinophils <0,15 at screening
* Signed informed consent

Exclusion Criteria:

* History of allergic asthma
* Doctor-diagnosed pneumonia within 6 weeks prior to screening
* Daily smoking or former daily smoking within the last 6 months
* Known other respiratory conditions such as COPD or pulmonary sarcoidosis
* Known other chronic conditions that could impact or prevent study participation, including severe heart conditions and conditions requiring treatment with immunosuppressive drugs such as Prednisolon, Methotrexate or biological treatments, assessed by study doctor
* Pregnancy or planned pregnancy
* Abuse of alcohol or other recreational drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-10-25 (Actual)

PRIMARY OUTCOMES:
Change in Control Questionnaire (ACQ) from baseline to post-tapered ICS | 52 weeks
Time from baseline to drop-out | 52 weeks

SECONDARY OUTCOMES:
Change in FeNO | 52 weeks
Change in FEV1 | 52 weeks
Change in blood eosinophils | 52 weeks
Change in serum periostin | 52 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Respiratory Research Unit, Copenhagen University Hospital Hvidovre, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mosbech CH, Godtfredsen NS, Ulrik CS, Westergaard CG. Biomarker-guided withdrawal of inhaled corticosteroids in asthma patients with a non-T2 inflammatory phenotype - a randomized controlled trial study protocol. BMC Pulm Med. 2023 Oct 4;23(1):372. doi: 10.1186/s12890-023-02679-y. PMID 37794472